CLINICAL TRIAL: NCT06515249
Title: Effectiveness and Safety of Integrative Therapies in Multiple Myeloma
Brief Title: Integrative Therapies in Multiple Myeloma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0054-24-BNZ
Record Dates: First submitted 2024-07-15; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Integrative Medicine; Quality-of-life; Complementary medicine; Hematology; Acupuncture; Mind-body; Touch
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrative medicine (Experimental): Integrative medicine treatments including acupuncture, touch, movement, mind-body, as patient's and staff's choice
  Interventions: Other: Integrative medicine
- Control (No Intervention)

INTERVENTIONS:
Other: Integrative medicine — Integrative medicine treatments including acupuncture, touch, movement, mind-body, as patient's and staff's choice
  Arms: Integrative medicine

SUMMARY:
Multiple myeloma is a hematologic malignancy that can cause anemia, renal failure, bone disease, and hypercalcemia. Today, myeloma is considered a chronic disease and most patients will receive ongoing biological treatments. As a result, this disease causes a number of symptoms related to the disease itself or its treatment, which include, among others, weakness and fatigue, bone or nerve pain, depression and anxiety, gastrointestinal symptoms, impairment of sexual function, etc. These symptoms cause significant damage to quality-of-life which is similar in patients who receive different treatment lines. As a result, the FDA emphasized quality-of-life as a key outcome for the approval of new drugs for the disease.

The conventional therapeutic approach to the various symptoms is based on supportive care guidelines including pharmacological and non-pharmacological treatment of pain, gastrointestinal symptoms, psychological components, etc. These treatments involve side effects and usually refer to individual symptoms.

Complementary and integrative medicine includes treatments of touch, movement, mind-body, acupuncture, nutrition and nutritional supplements. Many studies have shown the effectiveness of these treatments on various symptoms in cancer patients including pain, depression and anxiety, fatigue and weakness, gastrointestinal symptoms, etc. In myeloma patients, the effect of diet and nutritional supplements was mainly examined, but there is also little information on the effectiveness of mind-body treatments on symptoms of anxiety and depression, as well as acupuncture on neuropathy or on symptoms experienced by myeloma patients around autologous bone marrow transplantation.

In recent years, a wide variety of new drugs have entered the market that cause side effects that were unknown until now and little is known about the effect of complementary medicine treatments on symptoms and quality-of-life of myeloma patients since the development of these drugs.

In this study we will examine the effect of complementary and integrative medicine treatments (including acupuncture, touch, movement, mind-body) on the quality-of-life and symptoms that characterize myeloma patients during treatment with different lines of therapy, including new drugs.

Patients with a diagnosis of multiple myeloma who meet the study's inclusion criteria will be divided into the intervention group (complementary medicine treatments) and the control group (no treatments) according to their preferences. All the patients of the intervention group and the patients of the control group who agree will be asked to fill out quality-of-life questionnaires validated and translated into Hebrew, Arabic and Russian before the start of the treatment. The questionnaires include European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) which is a general quality-of-life questionnaire for cancer patients, with the addition of MY20 which is an addition of 20 specific questions for patients with multiple myeloma, the Edmonton Symptom Assessment System (ESAS) questionnaire which examines the severity of 10 common symptoms in patients with malignant disease, and the EuroQol-5 Dimension (EQ-5D) questionnaire which examines quality-of-life in cancer patients and is used as a primary outcome in many clinical studies. The same questionnaires will be sent again 1-2 weeks after the end of the treatments in the intervention group and 6-8 weeks after recruitment in the control group. Socio-demographic and medical data will also be collected from the patients and their medical records.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Diagnosis of multiple myeloma
* Possibility to answer questionnaires once a month in Hebrew, Arabic or Russian
* Signing an informed consent form

Exclusion Criteria:

* Age under 18 years
* In patients who will receive acupuncture: platelet level below 20x10^9/L
* In patients who will receive reflexology: deep vein thrombosis in the leg
* Hemodynamic instability
* Psychiatric disorder impairing competence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Quality-of-life specific to myeloma patients | From enrollment to 2 weeks after end of treatment in intervention group and 8 weeks after enrollment in control group
  EORTC QLQ-MY2 (European Organization for the Research and Treatment of Cancer Quality of Life for Myeloma patients) score at 1-2 weeks after end-of-treatment in intervention group and 7-8 weeks after recruitment in control group. It comprises 20 questions that address four myeloma-specific HRQoL domains: Disease Symptoms, Side Effects of Treatment, Future Perspective, and Body Image. Domain scores are averaged and transformed linearly to a score ranging from 0-100. A high score for Disease Symptoms and Side Effects of Treatment represents a high level of symptomatology or problems, whereas a high score for Future Perspective and Body Image represents better outcomes.

SECONDARY OUTCOMES:
General quality-of-life evaluation | From enrollment to 2 weeks after end of treatment in intervention group and 8 weeks after enrollment in control group
  European Organization Research for Treatment of cancer core quality of life (EORTC-QLQ-C30) questionnaire summary score which is calculated from the mean of 13 of the 15 quality-of-life (QLQ-C30) scales of the questionnaire = (Physical Functioning+ Role Functioning+ Social Functioning+ Emotional Functioning+ Cognitive Functioning+ 100-Fatigue+ 100-Pain+ 100-Nausea_Vomiting+ 100-Dyspnoea+ 100-Sleeping Disturbances+ 100-Appetite Loss+ 100-Constipation+ 100-Diarrhoea)/13. Scores range from minimum 0 to maximum 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
Symptom relief | From enrollment to 2 weeks after end of treatment in intervention group and 8 weeks after enrollment in control group
  Edmonton Symptom Assessment System (ESAS): assesses the severity over time of nine symptoms common among patients with cancer and other advanced illness: pain, tiredness, drowsiness, nausea, shortness of breath, appetite, depression, anxiety, and wellbeing. A higher score represents a higher ("worse") level of symptoms.
Compliance to conventional therapy | From enrollment to 1 year after enrollment
  Relative dose intensity (RDI) which is the ratio of delivered dose intensity (DDI) of myeloma treatment with standard dose intensity (SDI) of myeloma treatment = DDI/SDI
Economic analysis | From enrollment to 3 months after enrollment
  Calculation of quality-adjusted life years based on EuroQol-5 Dimension (EQ-5D) scale. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient indicates health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ visual analogue scale (VAS) records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Overall response rate (ORR) to myeloma treatment | From enrollment to 1 year after enrollment
  Percentage of patients who have a partial response or complete response to the treatment of myeloma
Progression-free survival (PFS) | From enrollment to 2 years after enrollment
  The length of time during and after the treatment of myeloma that patient lives and disease does not progress
Overall survival (OS) | From enrollment to 2 years after enrollment
  The length of time during and after the treatment of myeloma that patient lives

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Levy Yurkovski, MD, Principal Investigator — Bnai Zion Medical Center, Haifa, Israel
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT06515249/Prot_SAP_000.pdf